CLINICAL TRIAL: NCT03024034
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral TP-271 in Healthy Adult Subjects, Including 1 Cross-over Arm
Brief Title: A Phase 1 TP-271 Oral PK Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TP-271-003; 15-0061 (Other: NIAID)
Record Dates: First submitted 2017-01-09; First posted 2017-01-18 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — TP-271

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 25 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort B (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 50 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort C (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 100 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort D (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 150 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort E (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 200 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort F (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 300 mg single dose (n = 6) or matching placebo (n = 2)
  Interventions: Drug: TP-271
- Cohort G (Active Comparator): Oral dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 50 mg TP 271, cross-over to 50 mg TP 271/250 mg EDTA (n = 3); 50 mg TP 271/250 mg EDTA, cross-over to 50 mg TP 271 (n = 3); matching placebo, cross over to 250 mg EDTA (n= 1); or 250 mg EDTA, cross over to matching placebo (n = 1)
  Interventions: Drug: TP-271

INTERVENTIONS:
Drug: TP-271 — single oral dose of TP 271 or placebo, randomized 3:1, doses escalating as 25 mg, 50 mg, 100 mg, 150 mg, 200 mg, and 300 mg, and a final crossover cohort of 50 mg TP-271 and 50 mg TP-271 with 250 mg of EDTA, or placebo and 250 mg of EDTA

SUMMARY:
The purpose of this study is to determine the safety and tolerability of up to 6 different single ascending oral doses of TP-271, ranging from 25 mg to 300 mg, in healthy adult male or female subjects.

DETAILED DESCRIPTION:
This study is designed to assess oral TP-271, and the objectives of the study are to examine the safety, tolerability, and PK of oral TP-271 in healthy adult subjects after administration of a single dose. A single-dose, dose-escalating study design is common for early clinical studies. A cohort size of 8 subjects (6 receiving oral TP-271 and 2 receiving placebo) for the single ascending dose cohorts (Cohorts A through F) will allow sufficient data assessments of plasma and urine concentrations, plasma PK parameters, and safety without exposing large numbers of subjects to oral TP-271 in this clinical study. One additional cohort of 8 subjects will first receive treatment with TP-271 or TP-271 co-administered with ethylenediaminetetraacetic acid (EDTA) and then cross-over to treatment with the other study agent, which will allow a comparison of the bioavailability of TP-271 alone compared to TP-271 co-administered with EDTA, as well as allow additional assessment of plasma and urine concentrations, plasma PK parameters, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Be within the age range of 18 to 50 years, inclusive, at the time of Screening
2. Voluntarily sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved ICF to participate in the study after all relevant aspects of the study have been explained and discussed with the subject and before undergoing any study-related procedures
3. Have a body mass index (BMI) ≥18.0 and ≤33.0 kg/m2
4. Have a negative history of and negative screening results for human immunodeficiency virus 1 and 2 and hepatitis B and C antibodies
5. Have the ability to communicate with the study unit staff in a manner sufficient to carry out all protocol procedures as described
6. Female subjects must be of non-child bearing potential, either 1-year post menopausal or surgically sterile (bilateral oophorectomy, bilateral tubal ligation, or complete hysterectomy)
7. Male subjects must be willing and able to use a barrier method of contraception or practice abstinence (including male subjects who had a vasectomy) from dosing through 90 days post-dosing of the study drug

Exclusion Criteria:

1. History and/or presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal, endocrine, psychiatric, or mental disease or disorder, or mental or legal incapacitation, which, in the opinion of the PI, may either put the subject at risk because of participation in the study, influence the results of the study, or influence the subject's ability to participate in the study
2. Clinical laboratory values that fall outside the eligibility range specified in Appendix D are exclusionary; for laboratory values that are not included in Appendix D, values outside of the reference range are exclusionary with the following exceptions (Table 3):

   Table 3 Acceptable Out-of-Range Clinical Laboratory Values Low Chemistry Values High Chemistry Values Out-of-Range Urinalysis Values Out of Range Hematology Values Bicarbonate Chloride High or low specific gravity High hematocrit Chloride HDL cholesterol Cloudy Basophils GGT LDL cholesterol Mucus Monocytes HDL cholesterol Phosphorus Crystals MCV LDH Triglycerides Ketones MCHC LDL cholesterol Hyaline casts MCH Phosphorus High or low pH RBC Triglycerides Urobilinogen a Bicarbonate >18 mEq/L. b Ketonuria is acceptable only when the concurrent blood glucose is normal. c Measured when monitoring the serum bilirubin concentration. Abbreviations: GGT = gamma-glutamyltransferase; HDL = high-density lipoprotein; LDH = lactate dehydrogenase; LDL = low-density lipoprotein; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = mean corpuscular volume; RBC = red blood cell.
3. Known allergy to tetracycline antibiotics, EDTA, or any of the excipients in TP 271
4. Clinically significant abnormality on a 12-lead ECG including the following:

   * Rhythm other than sinus
   * Corrected QT interval using Fridericia's formula (QTcF) >450 msec
   * Evidence of second- or third-degree atrioventricular (AV) block
   * Pathological Q-waves (defined as a Q-wave >40 msec or depth >0.4 to 0.5 mV)
   * Evidence of ventricular pre-excitation
   * Evidence of complete left bundle branch block (BBB), right BBB, or incomplete left BBB
   * Intraventricular conduction delay with QRS duration >120 msec
   * ST segment abnormalities unless judged by the Investigator to be non pathologic
5. History of seizures
6. A history within 3 years of positive result on urine screen for drugs of abuse or a positive result at Screening for any of the following drugs of abuse: tetrahydrocannabinols, cocaine, opioids, phencyclidines, amphetamine, benzodiazepine, and barbiturates
7. Use of tobacco, nicotine, or nicotine-replacement products within 3 months prior to administration of study drug through the last study visit
8. Typical weekly alcohol consumption of 7 or more alcoholic drinks, where 1 alcoholic drink is defined as 1 glass of beer (approximately 10 to 12 oz), 1 can (12 oz) of beer, 1 glass of wine (approximately 4 to 5 oz), or distilled spirits (approximately 1 oz or 30 mL of liquor)
9. Alcohol consumption within 48 hours prior to dosing
10. Participation in a clinical study within 10 half-lives of the prior study treatment or within the previous 3 months (if the half-life of investigational agent is unknown) prior to receiving study drug on Day 1 or planned participation in another clinical study concurrent with the present trial
11. History of difficulty donating blood or poor venous access
12. Recent blood donation (1 unit or approximately 450 mL) within 1 month prior to receiving study drug or plans to donate prior to receiving study drug or during the clinical study
13. Use of any prescription or non-prescription medication, including vitamins or herbal medications, vaccination, or immunization within 7 days, or 5 half-lives (if known), whichever is longer, prior to dosing of study drug, with the following exceptions: medications used to treat an AE, and the use of acetaminophen, naproxen, and ibuprofen is permitted except for within 24 hours prior to dosing
14. Male subject donates or plans to donate sperm during the study and for at least 90 days after study drug administration.
15. Unwillingness or inability to follow the procedures outlined in the clinical study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Through study completion, approximately 39 days
  The incidence, intensity, and type of adverse events (AE) and the total number of participants experiencing AEs that are related to treatment
  Outcome measures to be collected in support of the primary objective (safety and tolerability) include:
  * The incidence, intensity, and type of AEs (from time of signing of informed consent form [ICF] through EOS);
  * Changes in physical examination findings (Day -1 and EOS);
  * Changes in vital signs (Day -1 through EOS);
  * Changes in safety laboratory (chemistry, hematology, coagulation, urinalysis) results (Days -1 through EOS); and
  * Changes in ECG measurements (Days -1 through EOS).
Physical Exams | Through study completion, approximately 39 days
  Changes in physical examination findings
Vital Signs | Through study completion, approximately 39 days
  Changes in vital signs
Safety Laboratory | Through study completion, approximately 39 days
  Changes in safety laboratory (chemistry, hematology, coagulation, urinalysis) results that are considered abnormal, clinically significant and related to treatment
ECG measurements | Through study completion, approximately 39 days
  Abnormal ECG measurements that are abnormal, clinically significant and related to treatment

SECONDARY OUTCOMES:
Plasma Pharmacokinetic (PK) Analysis | Days 1-5
  Plasma concentrations of TP-271 and its C-4 epimer TP-9555 for PK analysis
Urine Pharmacokinetic (PK) Analysis | Days 1-5
  Urine concentrations of TP-271 and its C-4 epimer TP-9555
PK parameters - Cmax | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Cmax [The maximum observed plasma concentration]
PK parameters - Tmax | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Tmax [The time from dosing at which Cmax is apparent]
PK parameters - C8 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C8 [The concentration at 8 hours post-dose]
PK parameters - C12 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C8 [The concentration at 8 hours post-dose]
PK parameters - C24 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C24 [The concentration at 24 hours post-dose]
PK parameters - AUC(0-last) | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC(0-inf) [The area under the concentration vs time curve from time zero extrapolated to infinity]
PK parameters - AUC(0-inf) | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC(0-inf) [The area under the concentration vs time curve from time zero extrapolated to infinity]
PK parameters - AUC% extrapolated | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC%extrapolated [The percentage of AUC(0-inf) accounted for by extrapolation]
PK parameters - Lambda-z | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Lambda-z [Slope of the regression line passing through the apparent elimination phase in a concentration vs time plot]
PK parameters - T1/2el | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for T1/2el [The elimination half-life]
PK parameters - CL | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for CL [Clearance: the volume of plasma cleared per unit time]
PK parameters - Vd | Days 1-5
  The PK parameters of the epimer/parent will be calculated for Cmax and AUC(0-inf).
PK parameters - epimer/parent | Days 1-5
  The PK parameters of the epimer/parent will be calculated for Cmax and AUC(0-inf).

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided